CLINICAL TRIAL: NCT01955733
Title: Safety and Efficacy of BI 695500 in Patients With Moderately to Severely Active Rheumatoid Arthritis: an Open-label Extension Trial
Brief Title: Safety and Efficacy of BI 695500 in Patients With Moderately to Severely Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Substance discontinued
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1301.4; 2013-002622-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-09-30; First posted 2013-10-07 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

ARMS (1):
- BI 695500 (Experimental): BI 695500, Two infusions separated by 2 weeks, Intravenous infusion
  Interventions: Drug: BI 695500

INTERVENTIONS:
Drug: BI 695500

SUMMARY:
The primary objective of this trial is to evaluate the long-term safety of BI 695500 in adult patients with moderately to severely active rheumatoid arthritis (RA) who have successfully completed treatment in Trial 1301.1.

ELIGIBILITY:
Inclusion criteria:

1. Must give written informed consent and be willing to follow this Clinical Trial Protocol.
2. Male or female patients, with moderately to severely active RA who have previously participated in the double-blind randomized clinical Trial 1301.1.
3. Current treatment for RA on an outpatient basis:

   1. Patients must continue to receive and tolerate oral or parenteral methotrexate (MTX) therapy at a dose of 15-25 mg per week (dose may be as low as 10 mg per week if the patient is unable to tolerate a higher dose).
   2. Patients must be willing to receive oral folic acid (at least 5 mg/week or as per local practice) or folinic acid (at least 1 mg per week or as per local practice) or equivalent during the entire trial.
   3. If receiving current treatment with oral corticosteroids (other than intra-articular or parenteral), the dose must not exceed 10 mg/day prednisolone or equivalent. During the 4 weeks prior to Baseline (Day 1) the dose must remain stable.
   4. Intra-articular and parenteral corticosteroids are not permitted throughout the trial, with the exception of IV administration of 100 mg methylprednisolone 30 to 60 minutes prior to each infusion as part of the trial procedures.
   5. Any concomitant non-steroidal anti-inflammatory drugs (NSAIDs) must be stable throughout the trial.
   6. Patients may be taking oral hydroxychloroquine provided that the dose is not greater than 400 mg/day, or chloroquine provided that the dose is not greater than 250 mg/day. These doses must have been stable for a minimum of 12 weeks prior to Day 1. The hydroxychloroquine or chloroquine treatment will need to be continued at a stable dose with the same formulation until the end of the trial.
4. For participants of reproductive potential (males and females), use of a medically acceptable method of contraception during the trial, i.e., a combination of 2 forms of effective contraception (defined as hormonal contraception, intrauterine device, condom with spermicide, etc.). Females of childbearing potential must also agree to use an acceptable method of contraception (see above) for 12 months following completion or discontinuation from the trial medication.

Exclusion criteria:

1. Patients receiving current treatment with corticosteroids must not be receiving a dose exceeding 10 mg/day prednisone or equivalent.
2. Serious underlying medical conditions, which, per the investigator¿s discretion, could impair the ability of the patient to participate in the trial (including but not limited to ongoing severe infection, severe immunosuppression, severe heart failure, uncontrolled hypertension, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease).
3. Pregnancy or breast feeding. For women of childbearing potential, a positive serum pregnancy test at the Screening Visit.
4. Patients who have significant cardiac disease, including but not limited to congestive heart failure of Class III or IV of the New York Heart Association (NYHA) classification; uncontrolled angina or arrhythmia; any uncontrolled or severe cardiovascular or cerebrovascular disease; or uncontrolled hypertension.
5. Treatment with IV or intramuscular corticosteroids. The only exception will be the administration of 100 mg IV methylprednisolone 30 to 60 minutes before each infusion as part of the trial procedures.
6. Any condition or treatment (including biologic therapies) that, in the opinion of the investigator, may place the patient at unacceptable risk during the trial.
7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times upper limit of normal (ULN).
8. Hemoglobin <8.0 g/dL.
9. Levels of Immunoglobulin G(IgG) <5.0 g/L.
10. Absolute neutrophil count <1500/µL.
11. Platelet count <75000/µL.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2016-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (43):
- United States (29):
  - 1301.4.5585 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1301.4.5727 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 1301.4.5725 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1301.4.5761 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1301.4.5765 Boehringer Ingelheim Investigational Site, El Cajon, California
  - 1301.4.5553 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 1301.4.5527 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1301.4.5771 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1301.4.5797 Boehringer Ingelheim Investigational Site, Santa Maria, California
  - 1301.4.5807 Boehringer Ingelheim Investigational Site, Upland, California
  - 1301.4.5809 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1301.4.5567 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1301.4.5561 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1301.4.5721 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1301.4.5811 Boehringer Ingelheim Investigational Site, Cumberland, Maryland
  - 1301.4.5507 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 1301.4.5715 Boehringer Ingelheim Investigational Site, Grand Rapids, Michigan
  - 1301.4.5787 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1301.4.5525 Boehringer Ingelheim Investigational Site, Toms River, New Jersey
  - 1301.4.5779 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1301.4.5717 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1301.4.5801 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1301.4.5549 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1301.4.5729 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1301.4.5757 Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 1301.4.5789 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 1301.4.5705 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1301.4.5597 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1301.4.5795 Boehringer Ingelheim Investigational Site, Beckley, West Virginia
- 1301.4.0303 Boehringer Ingelheim Investigational Site, Kortrijk, Belgium
- 1301.4.0609 Boehringer Ingelheim Investigational Site, Plovdiv, Bulgaria
- 1301.4.1705 Boehringer Ingelheim Investigational Site, Magdeburg, Germany
- 1301.4.1807 Boehringer Ingelheim Investigational Site, Athens, Greece
- 1301.4.3305 Boehringer Ingelheim Investigational Site, Sneek, Netherlands
- Poland (5):
  - 1301.4.3909 Boehringer Ingelheim Investigational Site, Bialystok
  - 1301.4.3907 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1301.4.3915 Boehringer Ingelheim Investigational Site, Krakow
  - 1301.4.3919 Boehringer Ingelheim Investigational Site, Warsaw
  - 1301.4.3917 Boehringer Ingelheim Investigational Site, Wroclaw
- Portugal (2):
  - 1301.4.4013 Boehringer Ingelheim Investigational Site, Amadora
  - 1301.4.4007 Boehringer Ingelheim Investigational Site, Lisbon
- Spain (2):
  - 1301.4.4809 Boehringer Ingelheim Investigational Site, Seville
  - 1301.4.4813 Boehringer Ingelheim Investigational Site, Seville

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 97 subjects were screened for eligibility to participate in this extension trial. 91 subjects met all inclusion and exclusion criteria and were assigned to receive treatment.
Groups:
- BI 695500: The subjects were administered BI 695500, concentrate for solution for infusion, 10 mg/mL by intravenous infusion. Two 1000 mg infusions were separated by 2 weeks.
  Each patient was treated with BI 695500 on Days 1 and 15, with a possible further two infusions at Weeks 24 and 26 for eligible responders.
- Rituxan From 1301.1: The Rituxan from 1301.1 recommended dose for use in patients with Rheumatoid Arthritis is 1000 mg by IV infusion followed by a second 1000 mg IV infusion 2 weeks later.
- MabThera From 1301.1: The MabThera from 1301.1 recommended dose for use in patients with Rheumatoid Arthritis is 1000 mg by IV infusion followed by a second 1000 mg IV infusion 2 weeks later.
Period: Period 1
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Started | 33 | 29 | 29
Completed | 32 | 29 | 29
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Period 2
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Started | 32 | 29 | 29
Completed | 20 | 10 | 8
Not Completed | 12 | 19 | 21
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2
Not completed — Study terminated by sponsor | 8 | 14 | 16
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Other not defined above | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Randomized Analysis Set [SAFRD]: All subjects randomized in 1301.1 [excluding open-label safety run-in subjects of trial 1301.1] who receive at least one dose of trial medication and subjects will be classified according to treatment received in trial 1301.1.
  2 subjects from 1301.1 safety run-in also received treatment in 1301.4, thus 88.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1 | Total
Number analyzed (Participants) | 30 | 29 | 29 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (11.23) | 56.3 (11.02) | 56.8 (8.95) | 55.9 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 22 | 67
  Male | 9 | 5 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Drug Related Adverse Events During the Treatment Phase
Description: This outcome measure presents percentage of patients with drug related adverse events during the treatment phase. Treatment Emergent Adverse Events (TEAEs) were defined as Adverse Events (AEs) that started or worsened in severity on or after the first dose of trial medication in this extension study [1301.4] and prior to the last date of trial medication + 180 days [inclusive]. Drug-related events were those considered by the investigator to have a causal relationship to trial medication.
Time Frame: Week 48
Population: Safety Randomized Analysis Set (SAFRD): All subjects randomized in 1301.1 [excluding open-label safety run-in subjects of trial 1301.1] who receive at least one dose of trial medication and subjects will be classified according to treatment received in trial 1301.1. 2 subjects from 1301.1 safety run-in also received treatment in 1301.4, thus 88.
Measure: Number; unit: Percentage of patients
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Number analyzed (Participants) | 30 | 29 | 29
Percentage of patients | 16.7 | 6.9 | 3.4

2. Secondary Outcome: Change From Baseline in Clinical Trial 1301.1 in Disease Activity Score 28 (DAS28) (Erythrocyte Sedimentation Rate [ESR]) at Week 48 of Clinical Trial 1301.4
Description: DAS-28 (ESR)** is an index containing a 28-joint count for tenderness (TJC28), 28 joint count for swelling (SJC28), natural logarithm of ESR (inflammation) (Ln[ESR]) and a general health component (GH) which is the patient's global assessment of disease activity and was used to describe the severity of RA. The DAS28 (ESR) Score is calculated as:
  DAS28(ESR) = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.70*ln(ESR) + 0.014*(GH). DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity. A clinically important change in DAS28 score is defined as an improvement in DAS28 score of at least 1.2.
  The mean change from baseline (in clinical trial 1301.1) at Week 48 in the DAS28 (ESR) score is presented.
Time Frame: Baseline in clinical trial 1301.1 up to Week 48 in clinical trial 1301.4.
Population: The Full Analysis Set (FAS) consisted of all subjects from the randomised set of clinical trial 1301.1 who received at least one dose of trial medication and had data recorded for at least 1 DAS28 (ESR or C-reactive Protein [CRP]) or American College of Rheumatology 20% response criteria (ACR20).
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on Scale
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Number analyzed (Participants) | 30 | 26 | 28
Units on Scale | -2.0 [-2.70 to -1.33] | -2.0 [-2.66 to -1.38] | -1.6 [-2.42 to -0.88]

3. Secondary Outcome: The Percentage of Patients Meeting the ACR20 [Based on Improvement Since Baseline in Trial 1301.1] at Week 48 of Trial 1301.4
Description: A subject has an ACR20 response if all of the following occur:
  * a > 20% improvement in the swollen joint count (66 joints)
  * a > 20% improvement in the tender joint count (68 joints)
  * a > 20% improvement in at least 3 of the following assessments: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, patient's assessment of physical function, as measured by the Health Assessment Questionnaire - Disability Index, or Acute phase reactant (CRP).
  The number of subjects meeting the ACR20 response criteria at Week 48 is presented.
Time Frame: Baseline in clinical trial 1301.1 up to Week 48 in clinical trial 1301.4.
Population: The FAS consisted of all subjects from the randomised set of clinical trial 1301.1 who received at least one dose of trial medication and had data recorded for at least 1 DAS28 (ESR or CRP) or ACR20.
Measure: Number; unit: Percentage of patients
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Number analyzed (Participants) | 30 | 26 | 28
Percentage of patients | 3.7 | 4.3 | 4.0

4. Secondary Outcome: The Percentage of Patients Who Meet the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Definition of Remission [Based on Improvement Since Baseline in Trial 1301.1] at Week 48 of Trial 1301.4
Description: To meet the ACR/EULAR Remission criteria*, the subject needed to satisfy the following criteria:
  * TCJ (68 joints) < 1
  * SJC (66 joints) < 1
  * CRP < 1 milligrams per decilitre
  * patient global assessment < 10. The patient global assessment for the definition of ACR/EULAR Remission was defined with a visual analog scale in millimetres (0-100).** The number of subjects meeting the ACR/EULAR Remission definition at Week 48 is presented.
Time Frame: Baseline in clinical trial 1301.1 up to Week 48 in clinical trial 1301.4.
Population: The FAS consisted of all patients from the randomised set of clinical trial 1301.1 who received at least one dose of trial medication and had data recorded for at least 1 DAS28 (ESR or CRP) or ACR20.
Measure: Number; unit: Percentage of patients
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Number analyzed (Participants) | 30 | 26 | 28
Percentage of patients | 0.0 | 0.0 | 0.0

5. Secondary Outcome: The Percentage of Patients Who Meet the EULAR Response [Good Response, Moderate Response, or no Response] [Based on DAS28 Improvement Since Baseline in Trial 1301.1] at Week 48 of Trial 1301.4
Description: This outcome measure presents percentage of patients who meet the EULAR response [good response, moderate response, or no response] [based on DAS28 improvement since baseline in trial 1301.1] at Week 48 of trial 1301.4.
Time Frame: Week 48
Population: FAS. Subjects who did not complete Week 48 are not presented.
Measure: Number; unit: Percentage of patients
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Number analyzed (Participants) | 30 | 26 | 28
Percentage of patients
  Good response | 0.0 | 0.0 | 0.0
  Moderate response | 3.3 | 7.7 | 0.0
  No response | 13.3 | 15.4 | 14.3
  Missing | 43.3 | 15.4 | 14.3

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the first dose of study medication in this extension study [1301.4] and prior to the last date of study medication + 6 months [180 days].
Description: AEs are presented for the Safety Randomised Analysis Set (SAF) which consisted of all randomised subjects who received at least one dose of trial medication in this extension study [1301.4].
Arm/Group | BI 695500 | Rituxan From 1301.1 | MabThera From 1301.1
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/29 | 2/29
Other Adverse Events (participants affected / at risk) | 7/30 | 8/29 | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=30) | Rituxan From 1301.1 (N=29) | MabThera From 1301.1 (N=29)
Cellulitis (Infections and infestations) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral microangiopathy (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695500 (N=30) | Rituxan From 1301.1 (N=29) | MabThera From 1301.1 (N=29)
Sinusitis (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 2 | 4
Viral upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Further development of BI 695500 has been stopped and the program was therefore prematurely discontinued on 03Sep2015. The decision was made by the Sponsor based on a strategic review of company's product portfolio and not due to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.